Title: Study 3 Learning Verbs and Pronouns

NCT Number: NCT05193500

Document date: 1/6/2025

The objective of this study was to see whether autistic and non-autistic children comprehend verbs and pronouns when they are presented as relevant to the child (e.g., addressed to them) or neutral (e.g., overheard). For verbs, the method was a behavioral experiment in which children's learning was measured by their eye gaze to the intended target verb meaning. For pronouns, pronouns were presented as part of a game in which the child was either the addressee of the pronoun or was not, and the child's comprehension was tested. The method was a behavioral experiment in which children played a game live with two experimenters who either addressed the child or each other with the pronouns to refer to an object that belonged to one of the three players. Children's selection of an object was the measure of pronoun comprehension.

## For verbs:

The primary dependent variable reported here for verbs is the proportion of time children spend looking at the target object in each condition. Track loss data points (that is, data points on which the child's gaze could not be ascertained) are removed from analysis.

The primary statistical test for this data is a one-sample t-test of the mean target looking by participant after children hear the verb.

## For pronouns:

The primary dependent variable reported here for pronouns is the first object children select by touching or pointing it. Trials on which children did not respond are removed from analysis.

The primary statistical test for this data is a one-sample t-test of the mean target selection by participant after children hear the pronoun.